CLINICAL TRIAL: NCT05129904
Title: Precise Profiling of Liver Disease Patients With DPMAS Therapy, Treating Optimal Patients and Achieving Hard Endpoint: a Multicenter, Cluster-controlled Study (PADSTONE Study)
Brief Title: Precise Profiling of Liver Disease Patients With DPMAS Therapy, Treating Optimal Patients and Achieving Hard Endpoint (PADSTONE Study)
Acronym: PADSTONE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Nanchang University (Other); Tianjin Third Central Hospital (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Beijing YouAn Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); West China Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); The Ninth Hospital of Nanchang (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Taihe Hospital (Other); Beijing 302 Hospital (Other); Shanghai Public Health Clinical Center of Fudan University (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); Southwest Hospital, China (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Qilu Hospital of Shandong University (Other); Beijing Ditan Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Shanghai Public Health Clinical Center (Other Government); Shandong Provincial Hospital (Other Government); The First Hospital of Jilin University (Other); Sichuan Provincial People's Hospital (Other); Huashan Hospital (Other); People's Hospital of Anshun City of Guizhou Province (Other); LanZhou University (Other); General Hospital of Ningxia Medical University (Other); Second Xiangya Hospital of Central South University (Other); The First Hospital of Yunnan Province (Unknown); Chengdu Public Health Clinical Center (Unknown); Ruijin Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Shandong Provincial Clinical Center for Public Health (Unknown); Shandong First Medical University (Other); The Second Hospital of Shandong University (Other); Second Affiliated Hospital of Nanchang University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Hunan Provincial People's Hospital (Other); Union Hospital, Tongji Medical College (Unknown); Zhengzhou University Affiliated Luoyang Centre Hospital (Unknown); Hebei Medical University Third Hospital (Other); The Second Hospital of Hebei Medical University (Other); Hainan People's Hospital (Other); Zunyi Medical College (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Guangxi University of Traditional Chinese Medicine (Unknown); People's Hospital of Guangxi Zhuang Autonomous Region (Other); First People's Hospital of Foshan (Other); First Affiliated Hospital of Fujian Medical University (Other); Capital Medical University (Other); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jinjun Chen, Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: NFEC-2021-259
Record Dates: First submitted 2021-10-31; First posted 2021-11-22 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: DPMAS Therapy in Liver Disease Patients
Keywords: double plasma molecular absorption system; liver disease; acute-on-chronic liver failure; mortality
MeSH Terms: conditions — Liver Diseases; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine，stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Double plasma molecular absorption system treatment: Patients treat with DPMAS alone or in combination with plasma exchange
  Interventions: Other: Double plasma molecular absorption system
- Standard medical therapy: Patients with standard medical therapy except for DPMAS treatment or other artificial liver support system

INTERVENTIONS:
Other: Double plasma molecular absorption system — DPMAS is an extracorporeal procedure that combines two hemoperfusion machines. During the procedure, toxic plasma is separated and cleansed by perfusion over two absorbers, and the final cleansed plasma is then returned to patients. It does not require large volumes of plasma and nor does it bear the risk of plasma-associated allergic reaction or disease transmissions. DPMAS can attenuate the jaundice in a short term and decrease the bilirubin concentration, which then reduces the toxicities of bile acid and high levels of bilirubin on the hepatocytes
  Other Names: DPMAS treatment
  Groups: Double plasma molecular absorption system treatment

SUMMARY:
Acute-on-chronic liver failure (ACLF) is life-threaten syndrome in patients with chronic liver disease. In China, hepatitis B virus (HBV) is the main etiology of cirrhosis and HBV-ACLF is characterized by multiple organs failure (liver, coagulation and kidney, etc.) and associated with high risk of short-tern death. For the treatment of ACLF patients, recent studies investigated the efficiency of extracorporeal liver support, such as albumin dialysis, plasma exchange. However, the efficiencies remain unclear. Liver transplantation is the most efficient way to improve the survival of ACLF patients, especially for those patients with three or more organ failure.

More recently，an extracorporeal system which is called double plasma molecular absorption system (DPMAS) was applied for the treatment of ACLF patients. DPMAS is an extracorporeal procedure that combines two hemoperfusion machines. During the procedure, toxic plasma is separated and cleansed by perfusion over two absorbers, and the final cleansed plasma is then returned to patients. It does not require large volumes of plasma and nor does it bear the risk of plasma-associated allergic reaction or disease transmissions. PMAS can attenuate the jaundice in a short term and decrease the bilirubin concentration, which then reduces the toxicities of bile acid and high levels of bilirubin on the hepatocytes. Although DPMAS treatment is applied in the clinical practice for those patients with liver failure, it still lack of compelling evidence in terms of real efficiency.

Thus, in this prospective, multicenter and cluster-controlled study, the investigators aim to identify the optimal liver disease patients by using hard endpoints (short-term mortality and disease progression). Moreover, this study will collect biological samples, including plasma, urine and stool, to explore the precise profiling of ACLF patients with DPMAS therapy by multi-omics detection.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients
2. Age >18 years
3. Chronic liver disease regardless of the etiology
4. Total bilirubin ≥ 12mg/dl and INR ≥ 1.5

Exclusion Criteria:

1. with more than three organ failures (SOFA criteria);
2. the pregnant;
3. with severe non-hepatic disease (such as chronic obstructive pulmonary disease level IV, chronic kidney disease with end-stage renal failure, myocardial infarction within 3 months before admission); 4) human immunodeficiency virus (HIV) infection without treatment;

5) patients with unstable hemodynamics caused by infection or acute bleeding; 6) hospital stays <48 hours; 7) diagnosis of hepatocellular carcinoma during screening period; 8) for the DPMAS clusters: patients unwilling to receive DPMAS treatment alone or in combination with PE; 9) for the SMT clusters: patients plan to receive DPMAS therapy or other ALSS; 10) not suitable to participate in this study judging by researchers; 11) not sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1:
  Liver failure patients (Total bilirubin ≥ 12mg/dl and INR ≥ 1.5) treat with DPMAS alone or in combination with plasma exchange
  Cohort 2:
  Liver failure patients (Total bilirubin ≥ 12mg/dl and INR ≥ 1.5) with standard medical therapy except for DPMAS treatment or other artificial liver support system
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The rate of progression with 4 weeks | 4 weeks
  The progression of ACLF with 4 weeks
The 4-week transplant-free mortality | 4 weeks
  The 4-week transplant-free mortality

SECONDARY OUTCOMES:
The transplant-free mortality within 12 weeks | 12 weeks
  The transplant-free mortality within 12 weeks
The improvement of ACLF with 12 weeks | 12 weeks
  The improvement of ACLF with 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jinjun Chen, Doctor, Study Director — Nanfang Hospital, Sourthern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China